CLINICAL TRIAL: NCT06722443
Title: The Microbiome as a Modifiable and Predictive Factor in Obesity Treatment: Impact of Nutritional Intervention With Probiotics and Prebiotics.
Brief Title: Impact of Nutritional Intervention With Probiotics and Prebiotics on Obesity.
Acronym: MicoBeBioticos
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, Alba Rodriguez Nogales, Full professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Fundación Pública Andaluza par
Record Dates: First submitted 2024-11-22; First posted 2024-12-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight; Obesity, Morbid; Metabolic Syndrome
Keywords: microbiome; obesity; metabolic syndrome; probiotics; prebiotics; symbiotics
MeSH Terms: conditions — Obesity; Overweight; Obesity, Morbid; Metabolic Syndrome | interventions — Probiotics; Prebiotics; Synbiotics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo treated with 500 mg/capsule/day of maltodextrin
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Prebiotic; Dietary Supplement: Synbiotic
- Probiotic (Active Comparator): capsules with 10^9 CFU/ day of Limosilactobacillus fermentum CECT5716
  Interventions: Dietary Supplement: Prebiotic; Dietary Supplement: Synbiotic
- Prebiotic (Active Comparator): 500 mg/capsule/day of olive leaf extract, containing 35% oleuropein, an amount comparable to what could be consumed through daily intake of extra virgin olive oil.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Synbiotic
- Symbiotic (Active Comparator): A combination of prebiotic and probiotic at the same doses.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Treatment with capsules with 10^9 CFU/ day of Limosilactobacillus fermentum CECT5716 during 6 months
  Arms: Placebo; Prebiotic; Symbiotic
Dietary Supplement: Prebiotic — Treatment with capsules 500 mg/capsule/day of olive leaf extract, containing 35% oleuropein during 6 months
  Arms: Placebo; Probiotic; Symbiotic
Dietary Supplement: Synbiotic — A pill with a combination of prebiotic and probiotic at the same doses during 6 months
  Arms: Placebo; Prebiotic; Probiotic

SUMMARY:
Obesity is one of the most severe and prevalent non-communicable diseases worldwide, affecting an estimated one-third of the population in Spain. It is a multifactorial disease that, in extreme cases such as morbid obesity, can become highly disabling and is associated with significant morbidity and mortality. This is because it serves as a risk factor for numerous chronic diseases, including metabolic conditions (type 2 diabetes mellitus), cardiovascular diseases (hypertension, atherosclerosis, etc.), and even cancer.

The exact etiopathogenic mechanisms are not fully understood, but subclinical inflammation is considered to form the basis of the metabolic (diabetes) and cardiovascular (endothelial dysfunction, dyslipidemia, etc.) disturbances that almost invariably accompany obesity. Additionally, alterations in the composition of the gut microbiota, or dysbiosis, are now recognized as playing a key role in the pathogenesis of obesity. This makes the gut microbiota a highly attractive therapeutic target for both the prevention and treatment of obesity, including less severe forms and morbid obesity.

In this context, the use of probiotics or extracts with prebiotic properties represents a particularly interesting strategy against obesity, offering a combination of efficacy and safety for treating these patients. Consequently, the general objective is proposed to evaluate the impact of dietary interventions aimed at modulating dysbiosis through the administration of a probiotic (Lactobacillus fermentum CECT5716), a standardized olive leaf extract with prebiotic properties, or a synbiotic (a combination of the olive leaf extract and L. fermentum CECT5716) on the clinical response of patients with moderate or morbid obesity. This will include determining its relationship with the immuno-metabolic system and the characteristic cardiovascular complications of obesity.

Furthermore, the evaluation of these treatments in experimental models of obesity, including morbid obesity requiring surgery, is also proposed. These models will include trials involving fecal material transfer into germ-free mice. These results will add significant value to the project by advancing our understanding of the underlying mechanisms of the disease. This will aid in the establishment of new diagnostic, prognostic, and therapeutic biomarkers, which are of great interest in reducing the incidence and prevalence of this current obesity epidemic.

The estimated duration for completing the project is 12 months, with its conclusion anticipated by March 2024.

DETAILED DESCRIPTION:
Obesity: The Epidemic of the 21st Century and a Public Health Concern. Obesity is one of the most severe and prevalent non-communicable diseases of the 21st century, representing a global public health problem that affects all age groups. In Spain, it is estimated that over 39% of adults (aged 25-60) are overweight and 20% are obese, with Andalusia being one of the regions with the highest rates, which continue to rise. Obesity is a multifactorial, recurrent, and progressive disease associated with significant physical and psychological complications, as well as considerable morbidity and mortality. It is a key risk factor for numerous chronic conditions, including metabolic syndrome (type 2 diabetes mellitus, hypertension, dyslipidemia) and the associated elevated risk of cardiovascular diseases.

Moreover, obesity can increase the risk of other diseases, including digestive, respiratory, and joint disorders, as well as various types of cancer (esophagus, colon, pancreas, prostate, and breast). Although the pathogenic mechanisms underlying obesity are not fully elucidated, it is understood that obesity is linked to a state of chronic low-grade systemic inflammation. Dysregulated adipose tissue functionality in obese individuals leads to elevated free fatty acid levels and increased production of inflammatory cytokines, establishing a vicious cycle that promotes the hypertrophy and hyperplasia of adipocytes, hallmarks of obesity.

The excessive production of these mediators and their release into the bloodstream have a profound impact on other organs and systems, contributing to the metabolic (e.g., diabetes) and cardiovascular (e.g., endothelial dysfunction, atherosclerosis) alterations that almost invariably accompany obesity. Consequently, obesity is associated with reduced quality of life and has a significant negative socioeconomic impact. It is also a determinant of several "intermediate risk factors," leading to increased mortality and reduced life expectancy.

The treatment of obesity involves lifestyle and dietary changes, often supplemented by pharmacological therapy, including appetite suppressants and fat absorption inhibitors. However, these strategies may be insufficient, and for severe obesity (BMI >35) or morbid obesity (BMI >40), surgical intervention is often necessary. Bariatric surgery, despite its effectiveness in reducing metabolic and cardiovascular comorbidities and improving survival and quality of life, involves significant complications due to patient characteristics and high costs. Moreover, over the last 30 years, there has been a marked increase in the prevalence of morbid obesity and, consequently, a greater demand for bariatric surgery.

While surgery reduces comorbidities and enhances patient outcomes, its effects on the gut microbiota remain suboptimal. As such, specific dietary interventions before and/or after surgery are needed to improve microbial gene richness and ensure long-term metabolic health.

The Gut Microbiome as a Modifiable Factor in Obesity. Numerous studies have highlighted the critical role of the gut microbiome in the development and maintenance of obesity and its associated conditions. Research shows that the microbiome composition in lean individuals differs significantly from that in obese individuals, a condition known as dysbiosis. Obese individuals exhibit an increased Firmicutes/Bacteroidetes ratio, reduced microbial diversity, and enhanced energy extraction efficiency from food.

Dysbiosis is also associated with increased intestinal permeability, allowing bacterial components such as lipopolysaccharides (LPS) to enter systemic circulation, which promotes endotoxemia and exacerbates inflammation. This altered microbial composition is linked to increased production of short-chain fatty acids (SCFAs), particularly propionate, which may contribute to lipogenesis and gluconeogenesis.

Severe dysbiosis is observed in morbidly obese patients, characterized by drastic reductions in microbial richness, intensified systemic inflammation, and metabolic disturbances. Although bariatric surgery improves weight, metabolic markers, and microbial diversity, it does not restore microbiota richness to levels observed in lean individuals. Therefore, dietary interventions targeting microbial restoration are critical for post-surgical recovery and long-term health.

Modulation of the Microbiome in Obesity: Probiotics and Prebiotics. The selective modulation of the gut microbiome using probiotics and prebiotics has emerged as a promising therapy for obesity. Probiotics, defined as live microorganisms that confer health benefits when administered in adequate amounts, offer several advantages, including strengthening the intestinal barrier, immunomodulation, and restoring dysbiosis. Commonly used probiotics in obesity management include strains from the Lactobacillus and Bifidobacterium genera.

Studies in both animal models and humans have demonstrated that specific strains can reduce body weight, fat accumulation, lipid profiles, and inflammatory markers. However, the overall efficacy in humans has been modest, necessitating further research to identify optimal strains, dosages, and treatment durations.

Lactobacillus fermentum CECT5716 has shown immunomodulatory properties in experimental models of colitis and hypertension. Preliminary unpublished studies suggest that it can reduce weight gain and systemic inflammation in obesity models, likely by improving dysbiosis and intestinal barrier function.

Prebiotics, non-digestible dietary components that selectively stimulate beneficial gut bacteria, are also effective in obesity management. Phenolic compounds, such as oleuropein from olive leaves, have shown significant prebiotic potential, reducing fat deposition, improving lipid and glucose profiles, and mitigating inflammation and vascular dysfunction in animal studies.

The current project aims to evaluate the effects of dietary supplementation with L. fermentum CECT5716 or a standardized olive leaf extract, alone or in combination, on clinical outcomes in patients with moderate and morbid obesity. Specifically, it will assess their impact on dysbiosis, metabolic and cardiovascular health, and post-surgical recovery in morbidly obese patients. The intervention's effectiveness will be correlated with adherence to a Mediterranean diet. By integrating microbiomic and metabolomic analyses, the study seeks to establish a personalized treatment framework for obesity.

H1: L. fermentum CECT5716 and/or olive leaf extract supplementation reduces inflammation, metabolic disturbances, and cardiovascular complications in obesity.

H2: These interventions restore dysbiotic gut microbiota composition and function.

H3: Supplementation improves post-operative outcomes in morbidly obese patients.

H4: Combining probiotic and prebiotic interventions provides synergistic benefits, maximizing efficacy.

This project offers a comprehensive approach to addressing obesity through microbiome modulation, paving the way for innovative, personalized therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Obesity and Associated Comorbidities (Prediabetes, Diabetes, Dyslipidemia, Hypertension).

Exclusion Criteria:

* Antibiotic treatment.
* Pregnancy.
* Clinical diagnoses of Inflammatory bowel disease.
* Clinical diagnosis of Celiac disease
* Clinical diagnosis of Hematological pathologies.
* Clinical diagnosis of Autoimmune or immunodeficiency diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the composition of the intestinal microbiome using metagenomic analysis | From enrollment (T0) to the end of treatment (6 months(T6))
  Microbial DNA will be isolated from the intestinal contents (feces) of different groups at various time points (T0 and T6). Taxonomic group identification will be performed through metagenomic sequencing using the Nextera XT Library Preparation Kit (Illumina). Sequencing will be conducted on a NovaSeq-6000 platform. To analyze the microbiota taxonomy, the RAST platform will be used to classify reads into different amplicon sequence variants (ASVs). A dynamic threshold will be applied to filter out false or incorrect ASVs, eliminating those contributing less than 0.1% of the total sequence count. The ASVs table will then be normalized per sample using subsampling (or rarefaction) to a minimum read count. QIIME wrapper scripts (v1.9.1) will be employed to classify reads into taxonomic units and to identify taxa with differential abundance between groups.
Evaluation of the treatment using integrated data analysis | From enrollment (T0) to the end of treatment (6 months(T6))
  The data obtained from the different determinations conducted will be automated for integrated analysis. Variables will be normalized, and qualitative variables will be categorized.
  Integrated bioinformatics analysis will compare and functionally correlate nutritional data, omics data (microbiomics, metabolomics, and immunological profiles) with clinical phenotypes (obese and morbidly obese patients) and treatments (probiotic, prebiotic, and synbiotic).
  This analysis will be based on Bayesian methods, which provide a statistical framework enabling the probabilistic integration of information across multiple analysis steps. All data will be analyzed using R and GraphPad Prism (version 8.4.1). This approach will allow the identification of relationships between microbiota impact and the administered treatments, as well as determine which treatment demonstrated the highest efficacy.

SECONDARY OUTCOMES:
Evaluation of serological biochemical profile | From enrollment to the end of treatment (6 months)
  In blood samples collected at different points of the study (baseline and endpoint), the following parameters will be assessed using an autoanalyzer (Beckman Coulter AU5800): serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and γ-glutamyl transpeptidase (GGT), total bilirubin, creatinine, uric acid, and lipid profile, including triglycerides (TG), total cholesterol (TC), high-density lipoprotein cholesterol (HDL), and low-density lipoprotein cholesterol (LDL). Serum leptin, IL-6, and TNF-α will be measured using the MILLIPLEX MAG Human Adipokine Magnetic Bead Panel (Millipore). Serum adiponectin, lipopolysaccharide-binding protein (LBP), and insulin will be quantified using ELISA kits. All variables will be quantified in IU/L.
Determination of the treatment impact on the metabolome profile | From enrollment (T0) to the end of treatment (6 months(T6))
  Metabolomic studies from serum samples at two different points (initial and final point) will be performed usign HPLC-GS-GC (min and m/z).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigacion Biomedica, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Sojo MJ, Ruiz-Malagon AJ, Hidalgo-Garcia L, Molina-Tijeras JA, Diez-Echave P, Lopez-Escanez L, Rosati L, Gonzalez-Lozano E, Cenis-Cifuentes L, Garcia-Garcia J, Garcia F, Robles-Vera I, Romero M, Duarte J, Cenis JL, Lozano-Perez AA, Galvez J, Rodriguez-Cabezas ME, Rodriguez-Nogales A. The Prebiotic Effects of an Extract with Antioxidant Properties from Morus alba L. Contribute to Ameliorate High-Fat Diet-Induced Obesity in Mice. Antioxidants (Basel). 2023 Apr 21;12(4):978. doi: 10.3390/antiox12040978. PMID 37107352
- [Background] Diez-Echave P, Vezza T, Algieri F, Ruiz-Malagon AJ, Hidalgo-Garcia L, Garcia F, Moron R, Sanchez M, Toral M, Romero M, Duarte J, Garrido-Mesa J, Rodriguez-Cabezas ME, Rodriguez-Nogales A, Galvez J. The melatonergic agonist agomelatine ameliorates high fat diet-induced obesity in mice through the modulation of the gut microbiome. Biomed Pharmacother. 2022 Sep;153:113445. doi: 10.1016/j.biopha.2022.113445. Epub 2022 Jul 22. PMID 36076560
- [Background] Molina-Tijeras JA, Diez-Echave P, Vezza T, Hidalgo-Garcia L, Ruiz-Malagon AJ, Rodriguez-Sojo MJ, Romero M, Robles-Vera I, Garcia F, Plaza-Diaz J, Olivares M, Duarte J, Rodriguez-Cabezas ME, Rodriguez-Nogales A, Galvez J. Lactobacillus fermentum CECT5716 ameliorates high fat diet-induced obesity in mice through modulation of gut microbiota dysbiosis. Pharmacol Res. 2021 May;167:105471. doi: 10.1016/j.phrs.2021.105471. Epub 2021 Jan 30. PMID 33529749
- [Background] Vezza T, Rodriguez-Nogales A, Algieri F, Garrido-Mesa J, Romero M, Sanchez M, Toral M, Martin-Garcia B, Gomez-Caravaca AM, Arraez-Roman D, Segura-Carretero A, Micol V, Garcia F, Utrilla MP, Duarte J, Rodriguez-Cabezas ME, Galvez J. The metabolic and vascular protective effects of olive (Olea europaea L.) leaf extract in diet-induced obesity in mice are related to the amelioration of gut microbiota dysbiosis and to its immunomodulatory properties. Pharmacol Res. 2019 Dec;150:104487. doi: 10.1016/j.phrs.2019.104487. Epub 2019 Oct 11. PMID 31610229